CLINICAL TRIAL: NCT04594941
Title: A Descriptive, Comparative, Randomized, Crossover Study of Flurpiridaz (18F) Injection for Positron Emission Tomography (PET) Imaging for Assessment of Myocardial Perfusion Imaging Quality Using High Performance Liquid Chromatography (HPLC) and Solid Phase Extraction (SPE) Manufacturing Processes
Brief Title: A Study of Flurpiridaz (18F) Injection for PET Imaging for Assessment of MPI Quality Using HPLC and SPE Manufacturing Processes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: GE-265-001
Record Dates: First submitted 2020-09-29; First posted 2020-10-20 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence: SPE-SPE (Experimental): Participants received 2 intravenous (IV) boluses of Flurpiridaz (18F) Injection manufactured by SPE process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 millicurie (mCi) (63 to 93 megabecquerel [MBq]) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
  Interventions: Drug: Flurpiridaz (18F) Injection
- Treatment Sequence: HPLC-HPLC (Experimental): Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by HPLC process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
  Interventions: Drug: Flurpiridaz (18F) Injection
- Treatment Sequence: SPE-HPLC (Experimental): Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by 2 different processes (1 dose manufactured by SPE followed by 1 dose manufactured by HPLC) at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
  Interventions: Drug: Flurpiridaz (18F) Injection
- Treatment Sequence: HPLC-SPE (Experimental): Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by 2 different processes (1 dose manufactured by HPLC followed by 1 dose manufactured by SPE) at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
  Interventions: Drug: Flurpiridaz (18F) Injection

INTERVENTIONS:
Drug: Flurpiridaz (18F) Injection — All participants received 2 IV boluses of Flurpiridaz (18F) Injection in a large peripheral vein at rest.

SUMMARY:
This was a Phase 2 prospective, randomized, crossover study of Flurpiridaz (18F) Injection for PET-MPI in participants referred for evaluation of known coronary artery disease (CAD) or for suspected CAD with intermediate to high pre-test probability (PTP). The objective is to assess the difference and variability between 2 sets of rest images synthesized by the same or 2 different manufacturing processes. Twenty-eight evaluable [participants were enrolled in this study and underwent 2 Flurpiridaz (18F) Injection PET-MPI at rest. Each participant attended a Screening Visit at least 2 days and up to 14 days prior to the first Flurpiridaz (18F) Injection PET-MPI. The participants were randomized 1:1:1:1 to 4 possible sequences of receiving 2 doses of Flurpiridaz (18F) Injection: 2 groups of 7 participants received 2 Flurpiridaz (18F) Injection doses synthesized by the same manufacturing processes (either HPLC or SPE) and 2 groups of 7 subjects will receive 2 Flurpiridaz (18F) Injection doses synthesized by different manufacturing processes (1 dose by HPLC followed by 1 dose by SPE or 1 dose by SPE followed by 1 dose by HPLC). All participants were followed up by telephone for adverse events (AEs) and serious AEs (SAEs) at 24 (+8) hours following each Flurpiridaz (18F) Injection administration.

ELIGIBILITY:
Inclusion Criteria:

* * The participant was a man or woman ≥18 years of age

  * The participant was undergoing evaluation of known CAD or for suspected CAD with an intermediate to high PTP.
  * The participant had read, signed, and dated an informed consent form (ICF) prior to any study procedures being performed, and was willing to allow the study investigator to make the participant's medical records available to GE Healthcare.
  * The participant was male or was a nonpregnant, nonlactating female who was either surgically sterile (had a documented bilateral tubal ligation and oophorectomy and/or documented hysterectomy [bilateral tubal ligation alone was insufficient]) or was post-menopausal (cessation of menses for more than 1 year); enrollment in the study without a pregnancy test at Screening was allowed for these categories of female participants. For women of childbearing potential, the results of either a urine or serum human chorionic gonadotropin pregnancy test (with the result known on the day of each radiopharmaceutical administration) must be negative. These participants must have been practicing appropriate birth control from the time of the screening to 30 days after the second radiopharmaceutical administration. Such methods included: hormonal contraception including oral contraceptives; intrauterine device; intrauterine hormone releasing system; bilateral tubal occlusion; vasectomized partner; sexual abstinence; adequate barrier method with spermicide (e.g., diaphragm, condom).
  * The participant was able and willing to comply with all study procedures as described in the protocol.

Exclusion Criteria:

* * Participants who were pregnant, may possibly be pregnant, or wish (including their partners) to become pregnant during the study period, or were lactating

  * Participants who were unable to undergo all of the imaging procedures
  * Participant with unstable cardiovascular condition, including but not limited to:

    1. Transient ischemic attack/stroke within 3 months of enrollment;
    2. Significant congenital heart disease;
    3. Uncontrolled hypertension;
    4. Uncontrolled tachyarrhythmia led to symptoms or hemodynamic compromise.
  * Participants required cardiac intervention (i.e., percutaneous coronary intervention or coronary artery bypass graft) before completing the study.
  * Primary hemodynamically significant uncorrected valvular heart disease, obstructive or regurgitant.
  * Participants with screening laboratory findings as follows:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) was greater than 3 times the upper limit of normal;
    2. Total bilirubin ≥2.0 mg/dL (34.2 μmol/L);
    3. Serum creatinine ≥3.0 mg/dL (265.2 μmol/L).
  * Participants who presented with any clinically active, serious, life-threatening disease, medical or psychiatric condition, and/or who have a life expectancy of <6 months, or for whom study participation may compromise their management; and participants whom the investigator judges to be unsuitable for participation in the study for any reason.
  * Participants undergone evaluation for heart transplantation or with a history of heart transplantation.
  * Participants enrolled in another clinical study within the 30 days before enrollment in this study.
  * Participants previously enrolled in this study or any Flurpiridaz (18F) Injection study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Tranquart, MD, PhD, Study Director — GE Healthcare
Locations (5):
- United States (5):
  - Indago Research and Health Center, Hialeah, Florida
  - Pioneer Clinical Studies, Miami, Florida
  - Amavita Clinical Research, LLC, North Miami Beach, Florida
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Memorial City and Katy Cardiology Associates, Katy, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 centers in the United States from 27 January 2022 and 26 May 2022.
Pre-assignment Details: A total of 38 participants were enrolled, of which 35 were randomized into 1 of 4 sequences: Solid phase extraction (SPE)-SPE, high performance liquid chromatography (HPLC)-HPLC, SPE-HPLC, HPLC-SPE) to receive either 2 doses of Flurpiridaz (18F) Injection manufactured by the same process (HPLC or SPE) or 2 doses manufactured by different processes (1 dose by HPLC and 1 dose by SPE in a random order).
Period: Overall Study
Arm/Group | Treatment Sequence: SPE-SPE | Treatment Sequence: HPLC-HPLC | Treatment Sequence: SPE-HPLC | Treatment Sequence: HPLC-SPE
Started | 7 | 10 | 11 | 7
Modified Intent-to-Treat (mITT) Population (mITT population included all participants who were randomized to receive >=1 dose of Flurpiridaz (18F) Injection and who completed the 2 rest Flurpiridaz (18F) Injection PET-MPI procedures.) | 7 | 7 | 10 | 7
Completed | 7 | 7 | 10 | 7
Not Completed | 0 | 3 | 1 | 0
Not completed — Other | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Sequence: SPE-SPE: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by SPE process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence: SPE-SPE | Treatment Sequence: HPLC-HPLC | Treatment Sequence: SPE-HPLC | Treatment Sequence: HPLC-SPE | Total
Number analyzed (Participants) | 7 | 10 | 11 | 7 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.30) | 62.7 (8.71) | 66.0 (9.75) | 63.1 (10.30) | 64.8 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3 | 3 | 9
  Male | 4 | 10 | 8 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 7 | 5 | 22
  Not Hispanic or Latino | 1 | 6 | 4 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 1 | 5
  White | 6 | 7 | 11 | 6 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intra-reader Difference of Summed Rest Score (SRS) for Positron Emission Tomography (PET) Myocardial Perfusion Imaging (MPI)
Description: 3 qualified readers (independent from the study) performed independent reads of all MPI images, inclusive of standard 17-segment polar-maps of perfusion defects. Each reader scored the perfusion pattern in each segment (17 segments) using a 5-point scale score range from 0 to 4: Normal 0, Minimal, mild impairment of perfusion = 1, Moderate impairment of perfusion = 2, Significant impairment of perfusion = 3, No perfusion = 4. Higher score indicated = impairment of perfusion. SRS was calculated by summing individual scores from each of 17 segments to give an overall score between 0 and 68; a score of 0 indicates normal outcome and scores more than 0 indicate increasingly worse outcomes as the score increases. The summed score of the 17 segments SRS was used for analysis. Intra-reader difference of SRS for PET MPI was reported.
Time Frame: Up to 2 weeks
Population: Analysis was performed on mITT population. A participant received SPE in both periods was counted twice in SPE group and a participant received HPLC in both periods was counted twice in HPLC group, while a participant received both methods is counted once in each group.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Flurpiridaz (18F): SPE: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by SPE process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 millicurie (mCi) (63 to 93 megabecquerel [MBq]) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
- Flurpiridaz (18F): HPLC: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by HPLC process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
Arm/Group | Flurpiridaz (18F): SPE | Flurpiridaz (18F): HPLC
Number analyzed (Participants) | 31 | 31
score on a scale
  Median of Readers | 6.662 (1.818) | 6.513 (1.818)
  Reader 1 | 6.235 (1.846) | 6.219 (1.846)
  Reader 2 | 7.009 (2.056) | 6.256 (2.056)
  Reader 3 | 7.336 (1.831) | 7.246 (1.831)
Statistical Analysis 1: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; Median of Readers: SPE VS HPLC Analysis was based on Mixed model repeated measures (MMRM) model include the median SRS in each dosing period as the dependent variable, with manufacturing process, period, and dosing sequence as fixed effects, and participant nested within sequence as the random effect; Test type: Other; p = 0.8452, Mixed-effects model for repeated measure; Least Sqaure (LS) Mean Difference = -0.149, 90% CI 2-sided [-1.431 to 1.133], Standard Error of Mean 0.754
Statistical Analysis 2: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; SPE VS HPLC: Reader 1 Analysis was based on Mixed model repeated measures (MMRM) model include the median SRS in each dosing period as the dependent variable, with manufacturing process, period, and dosing sequence as fixed effects, and participant nested within sequence as the random effect; Test type: Other; p = 0.9890, Mixed-effects model for repeated measure; LS Mean Difference = -0.015, 90% CI 2-sided [-1.899 to 1.868], Standard Error of Mean 1.109
Statistical Analysis 3: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; Reader 2: SPE VS HPLC Reader 2: Analysis was based on Mixed model repeated measures (MMRM) model include the median SRS in each dosing period as the dependent variable, with manufacturing process, period, and dosing sequence as fixed effects, and participant nested within sequence as the random effect; Test type: Other; p = 0.3852, Mixed-effects model for repeated measure; LS Mean Difference = -0.753, 90% CI 2-sided [-2.204 to 0.698], Standard Error of Mean 0.854
Statistical Analysis 4: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; Reader 3: SPE VS HPLC Analysis was based on MMRM model include the median SRS in each dosing period as the dependent variable, with manufacturing process, period, and dosing sequence as fixed effects, and participant nested within sequence as the random effect; Test type: Other; p = 0.9260, Mixed-effects model for repeated measure; LS Mean Difference = -0.091, 90% CI 2-sided [-1.735 to 1.554], Standard Error of Mean 0.968

2. Primary Outcome: Intra-reader Difference of Summed Rest Percent (SR%) for PET MPI
Description: 3 qualified readers (independent from the study) performed independent reads of all MPI images, inclusive of standard 17-segment polar-maps of perfusion defects. Each reader scored the perfusion pattern in each segment (17 segments) using a 5-point scale score range from 0 to 4: Normal 0, Minimal, mild impairment of perfusion = 1, Moderate impairment of perfusion = 2, Significant impairment of perfusion = 3, No perfusion = 4. Higher score indicated = impairment of perfusion. SRS was calculated by summing individual scores from each of 17 segments to give an overall score between 0 and 68; a score of 0 indicates normal outcome and scores more than 0 indicate increasingly worse outcomes as the score increases. Summed score of the 17 segments SRS was used for analysis. SR% is calculated by dividing the SRS by a number corresponding to the SRS value indicating a deficit of 4 in every segment and then multiplying the result by 100. Intra-reader difference of SR% for PET MPI was reported.
Time Frame: Up to 2 weeks
Population: Analysis was performed on mITT population. A participant received SPE in both periods was counted twice in SPE group and a participant received HPLC in both periods was counted twice in HPLC group, while a participant received both methods was counted once in each group.
Measure: Least Squares Mean (Standard Error); unit: percentage of score
Groups:
- Flurpiridaz (18F): SPE: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by SPE process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
Arm/Group | Flurpiridaz (18F): SPE | Flurpiridaz (18F): HPLC
Number analyzed (Participants) | 31 | 31
percentage of score
  Median of Readers | 9.797 (2.673) | 9.578 (2.673)
  Reader 1 | 9.168 (2.714) | 9.146 (2.714)
  Reader 2 | 10.307 (3.023) | 9.200 (3.023)
  Reader 3 | 10.789 (2.692) | 10.655 (2.692)
Statistical Analysis 1: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.8452, Mixed-effects model for repeated measure; LS Mean Difference = -0.219, 90% CI 2-sided [-2.104 to 1.667], Standard Error of Mean 1.109
Statistical Analysis 2: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; Reader 1: SPE VS HPLC Analysis was based on Mixed model repeated measures (MMRM) model include the median SRS in each dosing period as the dependent variable, with manufacturing process, period, and dosing sequence as fixed effects, and participant nested within sequence as the random effect; Test type: Other; p = 0.9890, Mixed-effects model for repeated measure; Least Square Mean (LSM) Difference = -0.023, 90% CI 2-sided [-2.793 to 2.747], Standard Error of Mean 1.630
Statistical Analysis 3: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; Reader 2: SPE VS HPLC Analysis was based on Mixed model repeated measures (MMRM) model include the median SRS in each dosing period as the dependent variable, with manufacturing process, period, and dosing sequence as fixed effects, and participant nested within sequence as the random effect; Test type: Other; p = 0.3852, Mixed-effects model for repeated measure; LS Mean Difference = -1.107, 90% CI 2-sided [-3.241 to 1.027], Standard Error of Mean 1.256
Statistical Analysis 4: Comparison: Flurpiridaz (18F): SPE vs Flurpiridaz (18F): HPLC; Reader 3: SPE VS HPLC Analysis was based on Mixed model repeated measures (MMRM) model include the median SRS in each dosing period as the dependent variable, with manufacturing process, period, and dosing sequence as fixed effects, and participant nested within sequence as the random effect; Test type: Other; p = 0.9260, Mixed-effects model for repeated measure; LS Mean Difference = -0.133, 90% CI 2-sided [-2.552 to 2.285], Standard Error of Mean 1.424

3. Primary Outcome: Intra-reader Correlation of SRS for PET MPI: Pearson's Correlation
Description: 3 qualified readers (independent from the study) performed independent reads of all MPI images, inclusive of standard 17-segment polar-maps of perfusion defects. Each reader scored the perfusion pattern in each segment (17 segments) using a 5-point scale score range from 0 to 4: Normal 0, Minimal, mild impairment of perfusion = 1, Moderate impairment of perfusion = 2, Significant impairment of perfusion = 3, No perfusion = 4. Higher score indicated = impairment of perfusion. SRS was calculated by summing individual scores from each of 17 segments to give an overall score between 0 and 68; a score of 0 indicates normal outcome and scores more than 0 indicate increasingly worse outcomes as the score increases. The summed score of the 17 segments SRS was used for analysis. Intra-reader correlation of SRS for PET MPI assessed using Pearson's correlation was reported.
Time Frame: Up to 2 weeks
Population: Analysis was performed on mITT population. SPE vs. HPLC was either SPE followed by HPLC or HPLC followed by SPE as a treatment sequence. Here, "overall number of participants analyzed" was the number of participants in MITT population for each treatment group.
Measure: Number; unit: Correlation coefficient of score
Groups:
- Flurpiridaz (18F): SPE vs SPE: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by SPE process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
- Flurpiridaz (18F): HPLC vs HPLC: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by HPLC process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
- Flurpiridaz (18F): SPE vs. HPLC: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by different processes (1 dose by SPE followed by 1 dose by HPLC or 1 dose by HPLC followed by 1 dose by SPE) at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
Arm/Group | Flurpiridaz (18F): SPE vs SPE | Flurpiridaz (18F): HPLC vs HPLC | Flurpiridaz (18F): SPE vs. HPLC
Number analyzed (Participants) | 7 | 7 | 17
Correlation coefficient of score
  Reader 1 | 1.000 | 0.890 | 0.787
  Reader 2 | 0.997 | 0.905 | 0.881
  Reader 3 | 0.999 | 0.931 | 0.910
Statistical Analysis 1: Comparison: Flurpiridaz (18F): SPE vs SPE; Reader 1; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Flurpiridaz (18F): SPE vs SPE; Reader 2; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Flurpiridaz (18F): SPE vs SPE; Reader 3; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 4: Comparison: Flurpiridaz (18F): HPLC vs HPLC; Reader 1; Test type: Other; p = 0.0072, Wilcoxon Signed Rank Test
Statistical Analysis 5: Comparison: Flurpiridaz (18F): HPLC vs HPLC; Reader 2; Test type: Other; p = 0.0051, Wilcoxon Signed Rank Test
Statistical Analysis 6: Comparison: Flurpiridaz (18F): HPLC vs HPLC; Reader 3; Test type: Other; p = 0.0023, Wilcoxon Signed Rank Test
Statistical Analysis 7: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 1; Test type: Other; p = 0.0002, Wilcoxon Signed Rank Test
Statistical Analysis 8: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 2; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 9: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 3; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test

4. Primary Outcome: Intra-reader Correlation of SRS for PET MPI: Kendall's Tau-b
Description: 3 qualified readers (independent from the study) performed independent reads of all MPI images, inclusive of standard 17-segment polar-maps of perfusion defects. Each reader scored the perfusion pattern in each segment (17 segments) using a 5-point scale score range from 0 to 4: Normal 0, Minimal, mild impairment of perfusion = 1, Moderate impairment of perfusion = 2, Significant impairment of perfusion = 3, No perfusion = 4. Higher score indicated = impairment of perfusion. SRS was calculated by summing individual scores from each of 17 segments to give an overall score between 0 and 68; a score of 0 indicates normal outcome and scores more than 0 indicate increasingly worse outcomes as the score increases. The summed score of the 17 segments SRS was used for analysis. Intra-reader correlation of SRS for PET MPI assessed using Kendall's tau-b was reported.
Time Frame: Up to 2 weeks
Population: as for outcome 3
Measure: Number; unit: Correlation coefficient of score
Arm/Group | Flurpiridaz (18F): SPE vs SPE | Flurpiridaz (18F): HPLC vs HPLC | Flurpiridaz (18F): SPE vs. HPLC
Number analyzed (Participants) | 7 | 7 | 17
Correlation coefficient of score
  Reader 1 | 1.000 | 0.732 | 0.769
  Reader 2 | 0.856 | 0.872 | 0.869
  Reader 3 | 1.000 | 0.733 | 0.833
Statistical Analysis 1: Comparison: Flurpiridaz (18F): SPE vs SPE; Reader 1; Test type: Other; p = 0.0089, Wilcoxon Signed Rank Test
Statistical Analysis 2: Comparison: Flurpiridaz (18F): SPE vs SPE; Reader 2; Test type: Other; p = 0.0207, Wilcoxon Signed Rank Test
Statistical Analysis 3: Comparison: Flurpiridaz (18F): SPE vs SPE; Reader 3; Test type: Other; p = 0.0089, Wilcoxon Signed Rank Test
Statistical Analysis 4: Comparison: Flurpiridaz (18F): HPLC vs HPLC; Reader 1; Test type: Other; p = 0.732, Wilcoxon Signed Rank Test
Statistical Analysis 5: Comparison: Flurpiridaz (18F): HPLC vs HPLC; Reader 2; Test type: Other; p = 0.0083, Wilcoxon Signed Rank Test
Statistical Analysis 6: Comparison: Flurpiridaz (18F): HPLC vs HPLC; Reader 3; Test type: Other; p = 0.0412, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 1; Test type: Other; p = 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 8: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 2; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test
Statistical Analysis 9: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 3; Test type: Other; p < 0.0001, Wilcoxon Signed Rank Test

5. Secondary Outcome: Variability of the SRS After MPI Sessions Using 2 Flurpiridaz (18F) Injection Doses by the Same Process
Description: Variability of SRS was estimated by using the SD of the paired difference divided by square root of 2. SRS was used for myocardial perfusion defects examination. The independent reads of all MPI images were based on standard 17-segment polar-maps of perfusion defects. Each reader scored the perfusion pattern in each segment (17 segments) using a 5-point scale score range from 0 to 4: Normal 0, Minimal, mild impairment of perfusion = 1, Moderate impairment of perfusion = 2, Significant impairment of perfusion = 3, No perfusion = 4. Higher score indicated = impairment of perfusion. SRS was calculated by summing individual scores from each of 17 segments to give an overall score between 0 and 68; a score of 0 indicates normal outcome and scores more than 0 indicate increasingly worse outcomes as the score increases. Variability of the SRS after MPI sessions using 2 Flurpiridaz (18F) injection doses by the same process was reported.
Time Frame: Up to 2 weeks
Population: Analysis was performed on mITT population. Here, "overall number of participants analyzed" signifies the participants with non-missing values receiving 2 doses with the same manufacturing process (either SPE-SPE or HPLC-HPLC). A participant received SPE in both periods was counted twice in SPE group and a participant received HPLC in both periods was counted twice in HPLC group, while a participant received both methods was counted once in each group.
Measure: Number; unit: (units on a scale)/(square root 2)
Arm/Group | Flurpiridaz (18F): SPE vs SPE | Flurpiridaz (18F): HPLC vs HPLC
Number analyzed (Participants) | 7 | 7
(units on a scale)/(square root 2)
  Reader 1 | 0.35 | 3.20
  Reader 2 | 2.67 | 2.06
  Reader 3 | 1.07 | 3.67

6. Secondary Outcome: Percentage of Participants With Intra-Reader Agreement of the Detection of Ischemic Defect on PET-MPI at Rest Between 2 MPI Acquisitions Using 2 Flurpiridaz (18F) Injection Doses
Description: Percentage of participants with intra-reader agreement of the detected ischemic defect on PET-MPI was reported.
Time Frame: Up to 2 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Flurpiridaz (18F): SPE vs. SPE: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by SPE process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 millicurie (mCi) (63 to 93 megabecquerel [MBq]) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
- Flurpiridaz (18F): HPLC vs. HPLC: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by HPLC process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
Arm/Group | Flurpiridaz (18F): SPE vs. SPE | Flurpiridaz (18F): HPLC vs. HPLC | Flurpiridaz (18F): SPE vs. HPLC
Number analyzed (Participants) | 7 | 7 | 17
percentage of participants
  Reader 1 | 100.0 | 71.4 | 94.1
  Reader 2 | 85.7 | 100.0 | 94.1
  Reader 3 | 100.0 | 100.0 | 94.1
Statistical Analysis 1: Comparison: Flurpiridaz (18F): SPE vs. SPE; Reader 1; Test type: Other; Kappa Statistics = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 2: Comparison: Flurpiridaz (18F): SPE vs. SPE; Reader 2; Test type: Other; Kappa Statistics = 0.6957, 95% CI 2-sided [0.1696 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 3: Comparison: Flurpiridaz (18F): SPE vs. SPE; Reader 3; Test type: Other; Kappa Statistics = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 4: Comparison: Flurpiridaz (18F): HPLC vs. HPLC; Reader 1; Test type: Other; Kappa Statistics = 0.4615, 95% CI 2-sided [-0.0699 to 0.9930] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 5: Comparison: Flurpiridaz (18F): HPLC vs. HPLC; Reader 2; Test type: Other; Kappa Statistics = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 6: Comparison: Flurpiridaz (18F): HPLC vs. HPLC; Reader 3; Test type: Other; Kappa Statistics = 1.0000, 95% CI 2-sided [1.0000 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 7: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 1; Test type: Other; Kappa Statistics = 0.8811, 95% CI 2-sided [0.6567 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 8: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 2; Test type: Other; Kappa Statistics = 0.8828, 95% CI 2-sided [0.6614 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics
Statistical Analysis 9: Comparison: Flurpiridaz (18F): SPE vs. HPLC; Reader 3; Test type: Other; Kappa Statistics = 0.8811, 95% CI 2-sided [0.6567 to 1.0000] — Kappa statistics was assessed using Cohen's kappa statistics

7. Secondary Outcome: Difference Between the Perfusion Rest Scores for Each of the 17 Segments and Each Reader for 2 Flurpiridaz (18F) Injection Doses From Same and Different Manufacturing Process
Description: Perfusion rest score was used for myocardial perfusion defects examination. The independent reads of all MPI images were based on standard 17-segment polar-maps of perfusion defects. Each reader scored the perfusion pattern in each segment (17 segments) using a 5-point scale score range from 0 to 4: Normal: 0; Minimal, mild impairment of perfusion, ambiguous image: 1; Moderate impairment of perfusion: 2; Significant impairment of perfusion: 3, No perfusion: 4. Higher score indicates impairment. Mean of the paired difference between the perfusion rest scores from 2 manufacturing processes for each of the 17 segments and each reader for 2 Flurpiridaz (18F) injection doses from same and different manufacturing process was reported.
Time Frame: Up to 2 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Difference of scores
Groups:
- Flurpiridaz (18F): SPE vs HPLC: Participants received 2 IV boluses of Flurpiridaz (18F) Injection manufactured by different processes (1 dose by SPE followed by 1 dose by HPLC or 1 dose by HPLC followed by 1 dose by SPE) at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
Arm/Group | Flurpiridaz (18F): SPE vs SPE | Flurpiridaz (18F): HPLC vs HPLC | Flurpiridaz (18F): SPE vs HPLC
Number analyzed (Participants) | 7 | 7 | 17
Difference of scores
  Reader 1: Segment 1 - Basal Anterior | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | -0.118 [-0.367 to 0.132]
  Reader 1: Segment 2 - Basal Anteroseptal | 0.000 [0.000 to 0.000] | -0.286 [-0.985 to 0.413] | 0.059 [-0.227 to 0.345]
  Reader 1: Segment 3 - Basal Inferoseptal | 0.000 [0.000 to 0.000] | -0.714 [-1.874 to 0.445] | 0.059 [-0.162 to 0.279]
  Reader 1: Segment 4 - Basal Inferior | 0.000 [0.000 to 0.000] | 0.286 [-0.594 to 1.165] | 0.235 [-0.152 to 0.622]
  Reader 1: Segment 5 - Basal Inferolateral | 0.000 [0.000 to 0.000] | 0.714 [-0.669 to 2.098] | 0.000 [-0.182 to 0.182]
  Reader 1: Segment 6 - Basal Anterolateral | 0.000 [0.000 to 0.000] | -0.143 [-0.492 to 0.207] | -0.471 [-0.956 to 0.014]
  Reader 1: Segment 7 - Mid Anterior | 0.000 [0.000 to 0.000] | 0.143 [-0.207 to 0.492] | -0.235 [-0.577 to 0.106]
  Reader 1: Segment 8 - Mid Anteroseptal | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.059 [-0.280 to 0.397]
  Reader 1: Segment 9 - Mid Inferoseptal | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.059 [-0.227 to 0.345]
  Reader 1: Segment 10 - Mid Inferior | 0.000 [0.000 to 0.000] | 0.143 [-0.981 to 1.267] | 0.059 [-0.162 to 0.279]
  Reader 1: Segment 11 - Mid Inferolateral | 0.000 [0.000 to 0.000] | 0.571 [-0.827 to 1.970] | 0.118 [-0.132 to 0.367]
  Reader 1: Segment 12 - Mid Anterolateral | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | -0.059 [-0.521 to 0.404]
  Reader 1: Segment 13 - Apical Anterior | 0.143 [-0.207 to 0.492] | -0.143 [-0.492 to 0.207] | 0.412 [-0.071 to 0.895]
  Reader 1: Segment 14 - Apical Septal | 0.000 [0.000 to 0.000] | 0.143 [-0.689 to 0.975] | 0.059 [-0.066 to 0.184]
  Reader 1: Segment 15 - Apical Inferior | 0.000 [0.000 to 0.000] | -0.143 [-0.492 to 0.207] | -0.176 [-0.698 to 0.345]
  Reader 1: Segment 16 - Apical Lateral | 0.143 [-0.207 to 0.492] | 0.000 [0.000 to 0.000] | 0.000 [-0.406 to 0.406]
  Reader 1: Segment 17 - Apex | 0.000 [0.000 to 0.000] | 0.286 [-0.991 to 1.562] | 0.000 [-0.364 to 0.364]
  Reader 2: Segment 1 - Basal Anterior | -0.429 [-1.477 to 0.620] | 0.286 [-0.166 to 0.737] | -0.235 [-0.524 to 0.054]
  Reader 2: Segment 2 - Basal Anteroseptal | 0.000 [0.000 to 0.000] | 0.000 [-0.534 to 0.534] | -0.176 [-0.448 to 0.095]
  Reader 2: Segment 3 - Basal Inferoseptal | -0.143 [-0.492 to 0.207] | 0.286 [-0.594 to 1.165] | 0.059 [-0.162 to 0.279]
  Reader 2: Segment 4 - Basal Inferior | 0.000 [0.000 to 0.000] | 0.286 [-0.594 to 1.165] | -0.235 [-0.622 to 0.152]
  Reader 2: Segment 5 - Basal Inferolateral | 0.429 [-0.620 to 1.477] | 0.000 [-1.413 to 1.413] | 0.176 [-0.150 to 0.503]
  Reader 2: Segment 6 - Basal Anterolateral | 0.286 [-0.874 to 1.445] | -0.143 [-0.975 to 0.689] | 0.000 [-0.603 to 0.603]
  Reader 2: Segment 7 - Mid Anterior | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | -0.176 [-0.379 to 0.026]
  Reader 2: Segment 8 - Mid Anteroseptal | 0.000 [0.000 to 0.000] | -0.143 [-0.492 to 0.207] | -0.176 [-0.503 to 0.150]
  Reader 2: Segment 9 - Mid Inferoseptal | -0.143 [-0.492 to 0.207] | 0.000 [-0.534 to 0.534] | 0.059 [-0.227 to 0.345]
  Reader 2: Segment 10 - Mid Inferior | -0.143 [-0.492 to 0.207] | 0.143 [-0.495 to 0.781] | -0.294 [-0.801 to 0.212]
  Reader 2: Segment 11 - Mid Inferolateral | -0.143 [-0.492 to 0.207] | 0.143 [-0.495 to 0.781] | 0.000 [-0.182 to 0.182]
  Reader 2: Segment 12 - Mid Anterolateral | 0.429 [-0.620 to 1.477] | 0.143 [-0.207 to 0.492] | 0.235 [-0.264 to 0.734]
  Reader 2: Segment 13 - Apical Anterior | 0.571 [-0.827 to 1.970] | 0.000 [0.000 to 0.000] | -0.118 [-0.288 to 0.053]
  Reader 2: Segment 14 - Apical Septal | 0.000 [0.000 to 0.000] | 0.143 [-0.689 to 0.975] | 0.059 [-0.162 to 0.279]
  Reader 2: Segment 15 - Apical Inferior | 0.000 [0.000 to 0.000] | -0.143 [-0.781 to 0.495] | 0.176 [-0.533 to 0.886]
  Reader 2: Segment 16 - Apical Lateral | 0.143 [-0.689 to 0.975] | -0.286 [-0.985 to 0.413] | -0.176 [-0.698 to 0.345]
  Reader 2: Segment 17 - Apex | -0.143 [-0.492 to 0.207] | -0.571 [-1.620 to 0.477] | 0.118 [-0.191 to 0.426]
  Reader 3: Segment 1 - Basal Anterior | 0.000 [0.000 to 0.000] | 0.429 [-0.620 to 1.477] | -0.118 [-0.288 to 0.053]
  Reader 3: Segment 2 - Basal Anteroseptal | 0.000 [0.000 to 0.000] | 0.429 [-0.620 to 1.477] | 0.059 [-0.162 to 0.279]
  Reader 3: Segment 3 - Basal Inferoseptal | 0.000 [0.000 to 0.000] | 0.143 [-0.689 to 0.975] | -0.059 [-0.279 to 0.162]
  Reader 3: Segment 4 - Basal Inferior | 0.000 [0.000 to 0.000] | 0.286 [-0.413 to 0.985] | 0.059 [-0.066 to 0.184]
  Reader 3: Segment 5 - Basal Inferolateral | 0.000 [0.000 to 0.000] | -0.286 [-1.950 to 1.379] | 0.235 [-0.355 to 0.825]
  Reader 3: Segment 6 - Basal Anterolateral | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | -0.059 [-0.279 to 0.162]
  Reader 3: Segment 7 - Mid Anterior | 0.000 [0.000 to 0.000] | 0.286 [-0.413 to 0.985] | -0.118 [-0.288 to 0.053]
  Reader 3: Segment 8 - Mid Anteroseptal | 0.000 [0.000 to 0.000] | 0.143 [-0.207 to 0.492] | 0.118 [-0.284 to 0.519]
  Reader 3: Segment 9 - Mid Inferoseptal | -0.429 [-1.477 to 0.620] | 0.143 [-0.207 to 0.492] | -0.176 [-0.379 to 0.026]
  Reader 3: Segment 10 - Mid Inferior | 0.000 [0.000 to 0.000] | 0.429 [-0.299 to 1.156] | 0.176 [-0.095 to 0.448]
  Reader 3: Segment 11 - Mid Inferolateral | 0.000 [0.000 to 0.000] | 0.143 [-0.689 to 0.975] | 0.118 [-0.424 to 0.659]
  Reader 3: Segment 12 - Mid Anterolateral | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | -0.176 [-0.448 to 0.095]
  Reader 3: Segment 13 - Apical Anterior | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.118 [-0.132 to 0.367]
  Reader 3: Segment 14 - Apical Septal | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.176 [-0.095 to 0.448]
  Reader 3: Segment 15 - Apical Inferior | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.000 [-0.481 to 0.481]
  Reader 3: Segment 16 - Apical Lateral | -0.143 [-0.492 to 0.207] | 0.000 [0.000 to 0.000] | -0.118 [-0.559 to 0.323]
  Reader 3: Segment 17 - Apex | 0.000 [0.000 to 0.000] | 0.857 [-0.598 to 2.312] | -0.176 [-0.698 to 0.345]

8. Secondary Outcome: Difference in Standard Uptake Value (SUV) of Time-activity Curves (TACs) by Region After MPI Sessions Using 2 Flurpiridaz (18F) Injection Doses Synthesized by Same and 2 Different Manufacturing Processes
Description: Difference was calculated by (Mean SUV from the second injection - Mean SUV from the first injection). SUV was calculated as Decay Corrected Uptake (kBq/cc) / (Injected Dose [MBq] / Weight (kilogram [kg]). Difference in SUV of TACs by region after MPI sessions using 2 Flurpiridaz (18F) injection doses synthesized by same and 2 different manufacturing processes was reported.
Time Frame: Up to 2 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Flurpiridaz (18F): SPE vs SPE | Flurpiridaz (18F): HPLC vs HPLC | Flurpiridaz (18F): SPE vs HPLC
Number analyzed (Participants) | 7 | 7 | 17
percent
  Blood | 2.445 (1.3493) | 1.677 (0.6376) | 2.097 (1.2356)
  Liver | 1.208 (0.6282) | 0.994 (0.7682) | 1.635 (1.6405)
  Lung | 1.652 (0.8000) | 1.507 (1.3117) | 1.110 (1.2815)
  Basal Anterior | 1.218 (0.8081) | 1.418 (0.7167) | 2.390 (2.7086)
  Basal Anteroseptal | 1.587 (0.8049) | 1.432 (0.6574) | 2.747 (2.8378)
  Basal Inferoseptal | 1.839 (0.7109) | 1.490 (0.5679) | 2.439 (2.5590)
  Basal Inferior | 1.582 (0.6831) | 1.365 (0.8715) | 2.144 (2.3601)
  Basal Inferolateral | 1.429 (0.7059) | 1.467 (0.5900) | 2.187 (2.5969)
  Basal Anterolateral | 1.477 (0.6315) | 1.612 (0.7959) | 2.390 (2.7995)
  Mid Anterior | 1.715 (1.1142) | 1.322 (0.9838) | 2.409 (2.8687)
  Mid Anteroseptal | 1.882 (1.0797) | 1.235 (0.7855) | 2.450 (2.8654)
  Mid Inferoseptal | 2.085 (0.9045) | 1.538 (1.0105) | 2.330 (2.6850)
  Mid Inferior | 2.132 (0.9901) | 1.564 (1.3300) | 2.211 (2.6039)
  Mid Inferolateral | 1.815 (0.8898) | 1.387 (0.9522) | 2.511 (3.1065)
  Mid Anterolateral | 1.847 (0.9456) | 1.408 (1.1032) | 2.605 (3.2431)
  Apical Anterior | 1.641 (0.9567) | 0.897 (0.5750) | 2.286 (2.6271)
  Apical Septal | 1.669 (0.9274) | 1.382 (1.1146) | 2.014 (2.3986)
  Apical Inferior | 2.037 (0.7632) | 1.312 (0.9000) | 1.986 (2.1610)
  Apical Lateral | 1.675 (1.0117) | 1.094 (0.7583) | 2.434 (2.7838)
  Apex | 1.424 (0.7731) | 1.105 (0.8259) | 1.833 (1.9528)
  Left Anterior Descending Artery (LAD) | 1.357 (0.9189) | 1.065 (0.7425) | 2.102 (2.6262)
  Left Circumflex Artery (LCX) | 1.503 (0.7590) | 1.194 (0.5908) | 2.248 (2.9416)
  Right Coronary Artery (RCA) | 1.846 (0.7726) | 1.319 (0.8727) | 2.052 (2.4344)
  Whole Myocardium | 1.449 (0.7983) | 1.100 (0.7513) | 2.052 (2.7089)

9. Secondary Outcome: Relative Difference in SUV (5- to 15-minute Perfusion Image) of TACs by Region After MPI Sessions Using 2 Flurpiridaz (18F) Injection Doses Synthesized by Same and 2 Different Manufacturing Processes
Description: Relative difference was calculated as 100 (SUV1-SUV2) / (0.5*[SUV1 + SUV2]) and SUV was calculated as Decay Corrected Uptake (kBq/cc) / (Injected Dose [MBq] / Weight [kg]). Relative difference in SUV of TACs by region after MPI sessions using 2 Flurpiridaz (18F) injection doses synthesized by same and 2 different manufacturing processes was reported.
Time Frame: Up to 2 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Flurpiridaz (18F): SPE vs SPE | Flurpiridaz (18F): HPLC vs HPLC | Flurpiridaz (18F): SPE vs HPLC
Number analyzed (Participants) | 7 | 7 | 17
percent
  Blood | 0.738 (27.4693) | 2.500 (32.0112) | -12.260 (22.1399)
  Liver | 5.965 (25.5980) | -2.200 (21.7720) | -6.042 (24.0731)
  Lung | -2.647 (34.8133) | -10.949 (35.3666) | 9.030 (39.7082)
  Basal Anterior | -1.991 (10.5622) | -9.725 (17.1715) | 3.246 (13.6798)
  Basal Anteroseptal | 1.031 (10.6386) | -5.606 (20.6948) | -2.130 (16.5611)
  Basal Inferoseptal | 7.157 (18.2437) | -4.976 (19.2974) | 1.540 (16.5447)
  Basal Inferior | 3.199 (13.1457) | -12.323 (21.9242) | 0.060 (17.9617)
  Basal Inferolateral | 2.525 (14.1960) | -14.008 (22.3971) | -2.293 (15.4717)
  Basal Anterolateral | 0.007 (15.6644) | -11.312 (18.2771) | 6.782 (12.5498)
  Mid Anterior | 0.591 (17.8879) | -12.036 (16.6875) | 3.186 (12.8762)
  Mid Anteroseptal | 4.007 (15.5683) | -7.183 (13.6480) | 0.789 (13.9519)
  Mid Inferoseptal | 4.716 (17.7702) | -12.442 (23.8374) | -0.140 (14.7096)
  Mid Inferior | 8.081 (21.0838) | -14.493 (30.8501) | -0.601 (16.8102)
  Mid Inferolateral | 6.665 (15.4194) | -12.251 (21.7680) | -1.414 (18.0348)
  Mid Anterolateral | 3.024 (17.5448) | -10.975 (14.4678) | 2.994 (13.5190)
  Apical Anterior | 6.649 (18.1637) | -3.935 (10.0975) | 1.708 (12.9038)
  Apical Septal | 5.473 (17.0274) | -6.934 (18.1451) | 0.802 (13.5151)
  Apical Inferior | 1.624 (20.8841) | -8.174 (15.6239) | -2.135 (16.0488)
  Apical Lateral | 2.404 (15.9485) | -2.015 (12.7979) | 0.133 (17.6721)
  Apex | 5.073 (17.2269) | -0.038 (15.2867) | -2.059 (11.0612)
  Left Anterior Descending Artery (LAD) | 2.088 (13.6375) | -7.123 (13.8785) | 1.212 (12.2860)
  Left Circumflex Artery (LCX) | 2.883 (14.1203) | -8.554 (13.5718) | -0.344 (15.0979)
  Right Coronary Artery (RCA) | 3.205 (16.8800) | -9.506 (18.8804) | -0.584 (15.3095)
  Whole Myocardium | 2.818 (14.3881) | -8.226 (14.2067) | 0.577 (13.2035)

10. Secondary Outcome: Number of Participants Categorized Based on Intra-Reader Agreement of the Image Quality Score Between the 2 Sets of PET Images for 2 Flurpiridaz (18F) Injection Doses From Different Manufacturing Processes
Description: Image quality scoring was performed as following: SPE image was worse than HPLC image when the difference (SPE - HPLC) score was less than or equal (<=)-3. SPE image was slightly worse than HPTC image when the difference score was <=-1 and greater than (>)-3. SPE and HPLC images were the same when the difference score was >-1 and less than (<) 1. SPE image was slightly better when the difference score >=1 and <3. SPE image was better when the difference was >=3. Higher score indicates better outcomes. Number of participants categorized based on intra-reader agreement of the image quality score between the 2 Sets of PET images for 2 Flurpiridaz (18F) injection doses from different manufacturing processes was reported.
Time Frame: Up to 2 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Flurpiridaz (18F): SPE vs. HPLC
Number analyzed (Participants) | 17
Participants
  Perfusion Image Quality: Reader 1: SPE image was worse than HPLC image | 1
  Perfusion Image Quality: Reader 1: SPE image was slightly worse than HPLC image | 3
  Perfusion Image Quality: Reader 1: SPE and HPLC images were the same | 11
  Perfusion Image Quality: Reader 1: SPE image was slightly better than HPLC image | 2
  Perfusion Image Quality: Reader 1: SPE image was better than HPLC image | 0
  Perfusion Image Quality: Reader 2: SPE image was worse than HPLC image | 0
  Perfusion Image Quality: Reader 2: SPE image was slightly worse than HPLC image | 1
  Perfusion Image Quality: Reader 2: SPE and HPLC images were the same | 16
  Perfusion Image Quality: Reader 2: SPE image was slightly better than HPLC image | 0
  Perfusion Image Quality: Reader 2: SPE image was better than HPLC image | 0
  Perfusion Image Quality: Reader 3: SPE image was worse than HPLC image | 0
  Perfusion Image Quality: Reader 3: SPE image was slightly worse than HPLC image | 3
  Perfusion Image Quality: Reader 3: SPE and HPLC images were the same | 13
  Perfusion Image Quality: Reader 3: SPE image was slightly better than HPLC image | 1
  Perfusion Image Quality: Reader 3: SPE image was better than HPLC image | 0
  Gated Image Quality: Reader 1: SPE image was worse than HPLC image | 0
  Gated Image Quality: Reader 1: SPE image was slightly worse than HPLC image | 5
  Gated Image Quality: Reader 1: SPE and HPLC images were the same | 9
  Gated Image Quality: Reader 1: SPE image was slightly better than HPLC image | 3
  Gated Image Quality: Reader 1: SPE image was better than HPLC image | 0
  Gated Image Quality: Reader 2: SPE image was worse than HPLC image | 0
  Gated Image Quality: Reader 2: SPE image was slightly worse than HPLC image | 3
  Gated Image Quality: Reader 2: SPE and HPLC images were the same | 12
  Gated Image Quality: Reader 2: SPE image was slightly better than HPLC image | 2
  Gated Image Quality: Reader 2: SPE image was better than HPLC image | 0
  Gated Image Quality: Reader 3: SPE image was worse than HPLC image | 0
  Gated Image Quality: Reader 3: SPE image was slightly worse than HPLC image | 6
  Gated Image Quality: Reader 3: SPE and HPLC images were the same | 8
  Gated Image Quality: Reader 3: SPE image was slightly better than HPLC image | 3
  Gated Image Quality: Reader 3: SPE image was better than HPLC image | 0

11. Secondary Outcome: Number of Participants Categorized Based on Intra-Reader Agreement of the Image Quality Score Between the 2 Sets of PET Images for 2 Flurpiridaz (18F) Injection Doses From Same Manufacturing Processes
Description: Image quality scoring was performed as following: 2 images were the same when the absolute difference score was >=0 and <1. 2 images were slightly different when the absolute difference score >=1 and <3. 2 images were different when the absolute difference score >=3. Higher score indicates better outcomes. Number of participants categorized based on intra-reader agreement of the image quality score between the 2 sets of PET Images for 2 Flurpiridaz (18F) injection doses from same manufacturing processes was reported.
Time Frame: Up to 2 weeks
Population: Analysis was performed on mITT population. Here, "overall number of participants analyzed" was the number of participants in MITT population for each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Flurpiridaz (18F): SPE vs SPE | Flurpiridaz (18F): HPLC vs HPLC
Number analyzed (Participants) | 7 | 7
Participants
  Perfusion Image Quality: Reader 1: 2 images were the same | 4 | 3
  Perfusion Image Quality: Reader 1: 2 images were slightly different | 3 | 3
  Perfusion Image Quality: Reader 1: 2 images were different | 0 | 1
  Perfusion Image Quality: Reader 2: 2 images were the same | 7 | 7
  Perfusion Image Quality: Reader 2: 2 images were slightly different | 0 | 0
  Perfusion Image Quality: Reader 2: 2 images were different | 0 | 0
  Perfusion Image Quality: Reader 3: 2 images were the same | 5 | 5
  Perfusion Image Quality: Reader 3: 2 images were slightly different | 2 | 2
  Perfusion Image Quality: Reader 3: 2 images were different | 0 | 0
  Gated Image Quality: Reader 1: 2 images were the same | 4 | 4
  Gated Image Quality: Reader 1: 2 images were slightly different | 3 | 3
  Gated Image Quality: Reader 1: 2 images were different | 0 | 0
  Gated Image Quality: Reader 2: 2 images were the same | 6 | 6
  Gated Image Quality: Reader 2: 2 images were slightly different | 1 | 1
  Gated Image Quality: Reader 2: 2 images were different | 0 | 0
  Gated Image Quality: Reader 3: 2 images were the same | 6 | 3
  Gated Image Quality: Reader 3: 2 images were slightly different | 1 | 4
  Gated Image Quality: Reader 3: 2 images were different | 0 | 0

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: A TEAE was defined as an adverse events (AE) that occurred from the time of investigational medicinal product (IMP) administration through the end of the follow-up period for the corresponding dose. Any medication error, clinically significant vital signs, electrocardiograms (ECGs), hematology, clinical chemistry laboratory tests, and urinalysis values determined by investigator were reported as TEAEs. Number of participants with TEAEs and serious TEAEs were reported.
Time Frame: From screening up to end of follow up (up to 30 days)
Population: The Safety Population included all participants who received >=1 dose of Flurpiridaz (18F) Injection in the study. Here, "overall number of participants analyzed" signifies those participants who took either one dose of IMP (SPE/HPLC) or two doses.
Measure: Count of Participants; unit: Participants
Groups:
- Flurpiridaz (18F): SPE: Participants received either 1 or 2 IV boluses of Flurpiridaz (18F) Injection manufactured by SPE process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
- Flurpiridaz (18F): HPLC: Participants received either 1 or 2 IV boluses of Flurpiridaz (18F) Injection manufactured by HPLC process at Visit 1 and 2.
  The targeted dose to the body of Flurpiridaz (18F) Injection was to be in the range of 1.7 to 2.5 mCi (63 to 93 MBq) for each administration and not exceed a total of 6 mCi (222 MBq) for an individual participant.
Arm/Group | Flurpiridaz (18F): SPE | Flurpiridaz (18F): HPLC
Number analyzed (Participants) | 25 | 27
Participants
  TEAEs | 3 | 1
  Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening up to end of follow up (up to 30 days)
Description: The Safety Population included all participants who received >=1 dose of Flurpiridaz (18F) Injection in the study. Participants at risk signifies those participants who took either one dose of IMP (SPE/HPLC) or two doses.
Arm/Group | Flurpiridaz (18F): SPE | Flurpiridaz (18F): HPLC
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 3/25 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flurpiridaz (18F): SPE (N=25) | Flurpiridaz (18F): HPLC (N=27)
Vomiting (Gastrointestinal disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT04594941/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04594941/SAP_003.pdf